CLINICAL TRIAL: NCT05997979
Title: Analgesic Effectiveness of Capsaicin 8% Cutaneous Patch for the Treatment of Chronic Postsurgical or Post-traumatic Neuropathic Pain: a Randomized Placebo Controlled Study in Children Aged 12 to 17-y
Brief Title: Analgesic Effectiveness of Capsaicin 8% Cutaneous Patch in Children
Acronym: CAPSAPED
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 29BRC21.0184
Record Dates: First submitted 2023-07-25; First posted 2023-08-18 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Neuropathic Pain; Chronic Pain
Keywords: Neuropathic Pain; Pediatric; Capsaicin; Randomized clinical trial
MeSH Terms: conditions — Neuralgia; Chronic Pain | interventions — Capsaicin; Transdermal Patch; Bandages, Hydrocolloid

STUDY DESIGN:
Intervention Model Description: Multicentric randomized controlled superiority trial in parallel arms:
  * experimental arm : Capsaicin 8% cutaneous patch
  * control arm : Hydrocolloid dressing
Who Masked: Participant
Masking Description: There is no mock cutaneous patch available for capsaicin 8% cutaneous patch. So we have chosen hydrocolloid dressing for placebo since it has no known effect on neuropathic pain and the tolerability is expected as excellent.
  The patient should not be aware of the specific aspect of capsaicin 8% patch and the protocol of application will be exactly the same. This should keep the patient blinded for the study treatment.
  The nurse who applies the patch is unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QUTENZA (Active Comparator): The experimental product is QUTENZA®, a cutaneous patch which contains 179 mg of capsaicin (capsaicin 8%).The patch measures 14 cm x 20 cm.
  The second application takes place three months after the first application.
  Interventions: Drug: Capsaicin 8% patch
- Placebo (Placebo Comparator): The placebo comparator is a hydrocolloid dressing: COMFEEL PLUS TRANSPARENT, a medical device class IIb commercialized by Coloplast. The patch measures 15 cm x 15 cm.
  The second application takes place three months after the first application.
  Interventions: Device: Hydrocolloid dressing

INTERVENTIONS:
Drug: Capsaicin 8% patch — Patients will receive Capsaicin 8% patch at the inclusion of the study and three months later if it is necessary (persistant pain). Qutenza should be applied to intact, non-irritated, dry skin, and during 30 minutes for the feet or 60 minutes for other areas of the body.
  Other Names: QUTENZA®
  Arms: QUTENZA
Device: Hydrocolloid dressing — Patients will receive Hydrocolloid dressing at the inclusion of the study and three months later if it is necessary (persistant pain). Hydrocolloid dressing should be applied to intact, non-irritated, dry skin, and during 30 minutes for the feet or 60 minutes for other areas of the body.
  Other Names: COMFEEL PLUS TRANSPARENT
  Arms: Placebo

SUMMARY:
This study concerns children aged to 12 to 17-years with local chronic neuropathic pain after trauma or surgery.

It is a multicentric randomized controlled superiority trial in parallel arms :

* experimental arm: Capsaicin 8% cutaneous patch
* controlled arm : Hydrocolloid dressing

Treatment with capsaicin application is realized at baseline, and repeated 3 months after the first patch application if needed.

Tolerance is assessed during each application and by phone call in following days until stop of cold need.

Efficacy is assessed monthly by clinical consultation until the end of the study (month 4).

DETAILED DESCRIPTION:
Children aged to 12 to 17-years monitored in pediatric pain outpatient clinics in the designed investigation centers for a local chronic neuropathic pain lasting more than 2 months after trauma or surgery are proposed to participate the trial.

Children with persistant neuropathic pain (DN4 (Diagnostic Neuropathic Pain) > or = 3/7 ou DN4 >or = 4/10) despite oral treatment following recommendations for neuropathic pain may be enrolled in the study.

For children not very painful (NRS-11 (Numeric Rating Scale) < 7 and FDI (Functional Disability Inventory) < 30) and without any oral treatment for neuropathic pain, the study may be proposed as first line treatment.

If both the child and his/her parents accept the trial, he/she will be included in the study.

It is a multicentric randomized controlled superiority trial in parallel arms :

* experimental arm: Capsaicin 8% cutaneous patch
* controlled arm : Hydrocolloid dressing

At M0, take place : baseline evaluation, agreement consent signature, inclusion and randomization, as well as first treatment application either capsaicin cutaneous patch or hydrocolloid dressing.

, If needed, the treatment may be done twice with a second application three months later (M3).

Tolerance is assessed during each application and by phone call in following days until stop of cold need.

Efficacy is assessed monthly by clinical consultation until the end of the study 4 months later (M4).

ELIGIBILITY:
Inclusion Criteria:

* Children aged 12 to 17 years (lower age limit of 12 has been chosen to ensure NPSI full filling).
* Male or female.
* Persistent neuropathic pain more than 3 months after surgery or trauma despite treatment following recommendations.
* Neuropathic pain is defined as a DN4 score equal to or greater than 3/7 or 4/10, and localized in a nerve territory explained by the surgery or the trauma.
* Treatment, survey and follow up must be realized in an identified investigating center of the study
* For patients of childbearing potential: use of an adequate method of contraception* during the course of the study through 48 hours after the last patch application (girls of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to the first patch application).

  * Adequate contraception includes sexual abstinence, progestogen-only oral hormonal contraception, where inhibition of ovulation is not the primary mode of action, male or female condom with or without spermicide, cap, diaphragm or sponge with spermicide, combination of male condom with either cap, diaphragm or sponge with spermicide (double barrier methods)

Exclusion Criteria:

* Intellectual deficiency not allowing full filling of NPSI.
* Insufficient command of the French language to full fill NPSI and other evaluation tools.
* Parents' refusal of consent.
* Minor patients' opposition.
* Underlying neurological disease.
* Ongoing neurotoxic treatment.
* Already treated by capsaicin.
* Cutaneous lesion on pain area.
* Patient presenting a pain area on the face, above the hairline of the scalp, and/or in proximity to mucous membranes
* Hypersensitivity to the active substance or to any of the excipients listed in section 6.1 of Qutenza SmPC.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2026-04-05 (Estimated); Study Completion 2026-04-05 (Estimated)

PRIMARY OUTCOMES:
The change in Neuropathic Pain Symptom Inventory score (NPSI) | At baseline (day of the patch application) and 4 months after patch application
  The decrease in Neuropathic Pain Symptom Inventory score (NPSI) is evaluated before the first application (M0) of capsaicin or placebo and 4 months later (M4).
  NPSI (Neuropathic Pain Syndrome Inventory) is a questionnaire without support, score from 0 to 100, higher score is worse outcome.

SECONDARY OUTCOMES:
Adverse event monitoring | At day 0, day 1, day 2, day 3 after patch application
  Adverse event monitoring are collected during patch application and by phone calls in the following days.
Vital signs | At baseline, Month 1, Month 2, Month 3 and Month 4
  Cardiac frequency in Bpm
Vital signs | At baseline, Month 1, Month 2, Month 3 and Month 4
  Arterial pressure in mmHg
Dermal assessment | At baseline
  Dermal assessment is evaluated with question concerning the treated area (YES/NO)
Dermal assessment | Month 1, Month 2, Month 3 and Month 4
  Dermal assessment is evaluated with questions concerning the feel of the treated area (YES/NO)
Treatment related pain and use of analgesic medication | At baseline, day 1, day 2, Month 1, Month 2, Month 3 and Month 4
  Intake of analgesic medication (YES/NO)
Duration of patch application | During patch application : at baseline and at Month 3 if it is applicable
  Duration of patch application in minutes
Neuropathic Pain Symptom Inventory score (NPSI) | At baseline, Month 1, Month 2, Month 3 and Month 4
  Global score and subscores of NPSI (Neuropathic Pain Syndrome Inventory) questionnaire without support, score from 0 to 100, higher score is worse outcome
Functional disability evaluation (FDI) | At baseline, Month 1, Month 2, Month 3 and Month 4
  Global score of FDI (Functional Disability Inventory) questionnaire, score from 0 to 60, higher score is worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Philippe J LE MOINE, MD, Principal Investigator — CHU of Brest
Locations (10):
- France (10):
  - CHU d'Amiens, Amiens
  - CHU d'Angers, Angers
  - CHU de Bordeaux, Bordeaux
  - CHU de Brest, Brest
  - CHU de Nantes, Brest
  - CHU de Lyon, Lyon
  - CHU de Marseille, Marseille
  - CHU de Montpellier, Montpellier
  - CHU de Tours, Tours
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.